CLINICAL TRIAL: NCT00628329
Title: Vitamin A, Its Receptors and Asthma: Vitamin A Levels in Serum and Expression and Responsiveness of Vitamin A Receptors in Circulating Mononuclear Cells of Asthmatics
Brief Title: Vitamin A, Its Receptors and Asthma
Status: Withdrawn | Type: Observational
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Selina Gierer, D.O., Assistant Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 11213
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Asthma
Keywords: asthma, retinol, cis-retinoic acid
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum without DNA, cells with DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
We wish to understand the association of Vitamin A serum levels and Vitamin A receptor number and responsiveness in asthmatics. We believe that Vitamin A receptors may be less prevalent in asthmatics and their responsiveness decreased.

DETAILED DESCRIPTION:
We wish to define the association of asthma, vitamin A serum levels and vitamin A receptor number and responsiveness on circulating mononuclear cells. Asthma is a complex, heterogenous and often debilitating and potentially deadly disease. The causes for asthma are many, with susceptibility and resistance to treatment is poorly understood. Ultimately, looking at this disease from another angle such as the role of Vitamin A and/or receptors can help us learn more about the pathophysiology and treatment of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously diagnosed asthma on inhaled corticosteroids, systemic steroids and/or long acting beta agonist (for a period of 6 mo to 5 years)
* Age 18-64
* Male or female

Exclusion Criteria:

* Children under age 18
* Adults 65 or older
* Patients with COPD

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male or female Age 18-64
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Retinol levels in blood, flow cytometric study of the RXRRAR receptors before and after addition of ATRA, 9-cis-RA and steroid | 2-4 weeks after blood sample drawn

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Stechschulte, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States